CLINICAL TRIAL: NCT00442091
Title: Dandelion Juice in the Treatment of Dyshidrotic Hand Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Evy Paulsen, Consultant dermatologist, Ph.D., Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070010
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Vesicular Palmoplantar Eczema; Pompholyx
Keywords: Dandelion; herbal remedy; hand eczema; Compositae
MeSH Terms: conditions — Eczema, Dyshidrotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10 ml of dandelion juice twice daily (Other)
  Interventions: Drug: dandelion juice

INTERVENTIONS:
Drug: dandelion juice — 10 ml bid for 20-30 days

SUMMARY:
Dandelion juice has been used in herbal medicine for at least 1000 years. Vesicular hand eczema is a rare, but difficult to treat, type of hand eczema. One case report has shown that ingestion of dandelion juice could induce a beneficial effect on this type of eczema. The purpose of this study is to test whether this effect can be retrieved in other patients.

DETAILED DESCRIPTION:
Dandelion juice has been used in herbal medicine for at least 1000 years. One case report has shown a beneficial effect of this herbal remedy on dyshidrotic hand eczema, and the purpose of this pilot study is to test whether this effect can be retrieved in other patients.

The patients are recruited from our out-patient clinic. Only patients with negative patch tests to Compositae are offered treatment with dandelion juice for 20-30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with dyshidrotic eczema for at least 1 year and negative patch test reactions to Compositae (tested within the last 3 years) and normal renal and hepatic blood tests.

Exclusion Criteria:

* Treatment with systemic steroids or other immunosuppressive/-modulating drugs, including UV therapy, within the last 3 months.
* Pregnancy, lactation.
* Compositae contact allergy.
* Liver or gall bladder disease.
* Abnormal renal or hepatic blood tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Improvement in dyshidrotic hand eczema in the study period assessed by HECSI score. | 3-4 weeks

SECONDARY OUTCOMES:
Improvement in dyshidrotic eczema in the study period assessed by the patient (Visual Analog Scale). | 3-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Evy Paulsen, Dr., Principal Investigator — Department of Dermatology, Odense University Hospital, DK-5000 Odense C
Locations (1):
- Department of Dermatology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No